CLINICAL TRIAL: NCT02052128
Title: Phase 1-2 Study of Onapristone in Patients With Progesterone Receptor Expressing Cancers
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arno Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARN-AR18-CT-101
Record Dates: First submitted 2014-01-28; First posted 2014-01-31 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Progesterone Receptor Positive Tumor: Max 1 Line of Prior Chemotherapy, no Prior Hormone Therapy
Keywords: endometrial cancer; ovarian cancer; breast cancer; uterine sarcoma; uterine endometrioid adenocarcinoma
MeSH Terms: conditions — Endometrial Neoplasms; Ovarian Neoplasms; Breast Neoplasms | interventions — onapristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- onapristone 10 mg BID mg (Experimental): onapristone 10 mg BID extended-release tablets
  Interventions: Drug: onapristone
- onapristone 20 mg BID (Experimental): onapristone 20 mg BID extended-release tablets
  Interventions: Drug: onapristone
- onapristone 30 mg BID (Experimental): onapristone 30 mg BID extended-release tablets
  Interventions: Drug: onapristone
- onapristone 40 mg BID mg (Experimental): onapristone 40 mg BID mg extended-release tablets
  Interventions: Drug: onapristone
- onapristone 50 mg BID (Experimental): onapristone 50 mg BID extended-release tablets
  Interventions: Drug: onapristone
- onapristone 100 mg QD (Experimental): onapristone 100 mg QD immediate-release tablets
  Interventions: Drug: onapristone

INTERVENTIONS:
Drug: onapristone
  Other Names: ZK 98299

SUMMARY:
This is a multi-center, open-label, randomized, parallel group two-stage phase 1 study with a phase 2 expansion component in pts with recurrent or metastatic APRpos uterine endometrioid adenocarcinoma. Stage 1: Six dose cohorts, 5 using the extended release tablet (ER) formulation (10 mg BID, 20 mg BID, 30 mg BID, 40 mg BID, 50 mg BID) and 1 using the immediate-release (IR) tablet formulation 100 mg QD will be randomized in parallel. After enrollment of 36 patients in Stage 1, a dose of 50 mg BID was determined to be the RP2D. Stage 2: An additional 10 patients with recurrent or metastatic APRpos uterine endometrioid adenocarcinoma (Stage 2a) will be enrolled at the RP2D. Based on the response in Stage 2a, the cohort will be further expanded by up to 19 more patients to a total of 29 patients to confirm the efficacy and safety profile of onapristone in this selected patient population (Stage 2b).

ELIGIBILITY:
Inclusion Criteria:

1. Post- menopausal female patients, 18 years of age or greater.
2. In Stage 1, recurrent or metastatic PR-expressing cancer that has the potential to benefit from an anti-progestin treatment including but not limited to endometrial cancer, ovarian, or breast cancer or uterine sarcoma. In Stage 2, recurrent or metastatic PR-expression uterine endometrioid adenocarcinoma that is determined to be APRpos.
3. Patients who have metastatic or recurrent disease after previous surgery, radiation therapy, and/or chemotherapy are eligible. In Stage 1, no restriction is placed on the number of prior therapies. In Stage 2, patients may have 0 or 1 prior chemotherapy treatments for adjuvant or metastatic disease and no prior endocrine therapies.
4. In Stage 1, evaluable disease per RECIST 1.1. In Stage 2, measurable disease.
5. Appropriate archival OR current tissue blocks or biopsy specimens to determine ER/PR and APR status.
6. Signed, written informed consent must be obtained and documented according to ICH-GCP, the local regulatory requirements, and local data protection laws prior to study-specific screening procedures.
7. ECOG performance status 0-1.
8. Health care coverage.

Exclusion Criteria:

1. Calculated creatinine clearance of <60 mL/min in Stage 1 and <40 mL/min in Stage 2
2. Patients with any other prior malignancy are not allowed except for the following:

   * Adequately treated basal cell or squamous cell skin cancer
   * In situ cervical cancer
   * Adequately treated Stage I or II cancer from which the patient is currently in complete remission or other cancer from which the patient has been disease-free for 2 years
3. Body mass index (BMI) <18.5 or >35 kg/m2.
4. On ECG a QTc(F) interval >480 msec or any clinically significant cardiac rhythm abnormalities.
5. Liver function tests documented within the screening period and on day -1 of treatment period:

   * Total bilirubin > ULN (except in patients diagnosed with Gilbert's disease).
   * Alkaline phosphatase > UNL or > 2.5 x UNL in case of liver metastases, or > 5 x UNL in case of bone metastases.
   * ALT/AST > UNL or > 2.5 x UNL in case of liver metastases.
6. Known positive virology/serology for human immunodeficiency virus (HIV)-1, HIV-2, hepatitis B (surface antigen), or hepatitis C.
7. Chronic inflammatory liver condition.
8. Chronic adrenal failure or is receiving concurrent long-term corticosteroid therapy.
9. History or clinical evidence of any surgical or medical condition which the investigator judges as likely to interfere with the results of the study or pose an additional risk in participating.
10. Used any prescription medication during the prior 1 month that the investigator judges is likely to interfere with the study or to pose an additional risk to the patient in participating.
11. Received an investigational product or been treated with an investigational device within 30 days prior to first drug administration, or plans to start any other investigational product or device study within 30 days after last drug administration.
12. Received prior systemic anticancer treatment (chemotherapy, targeted therapies including kinase inhibitors, antibodies, etc) less than 5 half-lives before the first dose of study drug or radiotherapy within 30 days; toxicity of the anticancer treatment must have recovered to grade 1 or less.
13. Current progestin-based hormone replacement therapy.
14. Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to swallow pills.
15. Has a mental incapacity or language barriers precluding adequate understanding, co-operation, and compliance with the study requirements.
16. Is, in the judgment of the investigator, unable or unwilling to comply with the requirements of the study.
17. Uncontrolled brain metastases or treatment by neurosurgical resection or brain biopsy within 4 weeks prior to Day 1.
18. For Stage 2 only, mixed histology i.e. patients with >10% non-endometrioid malignant cells in provided histopathology samples.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-10 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Stage 1: RP2D of a single agent extended-release tablet formulation of oral onapristone for future clinical development. | Baseline to 57 days post-first dose
Stage 2: ORR using RECIST 1.1 in 10-29 patients with recurrent or metastatic uterine endometrioid adenocarcinoma that is APRpos, and to determine the relationship between APR status and onapristone anti-tumor activity. | Baseline to 30 Days after last dose

SECONDARY OUTCOMES:
Safety and tolerability of extended-release onapristone tablets BID and of immediate-release onapristone tablets QD | Baseline to 30 Days after last dose
  Safety will be assessed by physical exam, vital signs, monitoring of adverse events, changes in ECG, and other clinical laboratory values
Comparison of safety of extended-release BID vs. immediate release QD schedules | Baseline to 30 Days after last dose
  Safety will be assessed by physical exam, vital signs, monitoring of adverse events, changes in ECG, and other clinical laboratory values
Anti-tumor activity based on tumor assessments (RECIST 1.1) and dates of progression | Baseline to 30 Days after last dose
PK of onapristone, mono-demethylated onapristone and other metabolites in plasma and urine | Baseline to 30 Days after last dose
  AUC, Cmax, Tmax, t1/2

CONTACTS AND LOCATIONS:
Overall Officials: Paul H Cottu, MD, Principal Investigator — Institut Curie, Paris, France
Locations (3):
- France (3):
  - Centre Oscar Lambret, Lille
  - Institut Curie Oncologie Medicale, Paris
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Cottu PH, Bonneterre J, Varga A, Campone M, Leary A, Floquet A, Berton-Rigaud D, Sablin MP, Lesoin A, Rezai K, Lokiec FM, Lhomme C, Bosq J, Bexon AS, Gilles EM, Proniuk S, Dieras V, Jackson DM, Zukiwski A, Italiano A. Phase I study of onapristone, a type I antiprogestin, in female patients with previously treated recurrent or metastatic progesterone receptor-expressing cancers. PLoS One. 2018 Oct 10;13(10):e0204973. doi: 10.1371/journal.pone.0204973. eCollection 2018. PMID 30304013